CLINICAL TRIAL: NCT03141619
Title: Cerebral Oxygenation and Neurological Outcomes FOllowing CriticAL Illness-2
Acronym: CONFOCAL-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Gordon Boyd (Other)
Collaborators: University Health Network, Toronto (Other); Vancouver General Hospital (Other); Western University, Canada (Other); University of Ottawa (Other); Université de Montréal (Other); University of Calgary (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Dr. Gordon Boyd, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: CTO Project ID 0815
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Critical Illness; Respiratory Failure; Shock; Delirium
Keywords: cerebral oximetry; near-infrared spectroscopy; neurocognitive; post-ICU syndrome
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Shock; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be collected for proteomic assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Respiratory failure and/or shock: All enrolled patients will undergo 72 hours of monitoring of cerebral oxygenation with near-infrared spectroscopy.

SUMMARY:
This study is designed to test the hypothesis that poor cerebral perfusion during critical illness is a risk factor for acute and long-term neurological dysfunction among survivors. We use near-infrared spectroscopy to measure brain tissue oxygenation as a non-invasive surrogate marker for cerebral perfusion. Acute neurological dysfunction is defined as the presence of delirium, which is assessed using the Confusion Assessment Method-Intensive Care Unit (CAM-ICU). Chronic neurological dysfunction is defined as having quantitative impairments on robotic testing (KINARM robot) and traditional neuropsychological screening (Repeatable Battery for the Assessment of Neuropsychological Status).

ELIGIBILITY:
Inclusion

1. Adults ≥ 18 years old
2. Admitted to a critical care unit requiring one or more of the following:

   (a) Respiratory failure requiring invasive mechanical ventilation with an expected duration >24 hours (b) Shock of any etiology. Shock is defined by the need for one of the following vasopressors/inotropes: (i) Dopamine ≥7.5 mcg/kg/min (ii) Dobutamine ≥5 mcg/kg/min (iii) Norepinephrine ≥5 mcg/min (iv) Phenylephrine ≥75 mcg/min (v) Epinephrine at any dose (vi) Milrinone at any dose (if used in conjunction with another agent) (vii) Vasopressin ≥0.03 u/min(if used in conjunction with another agent)

Exclusion:

1. Admission to the ICU > 24 hours
2. Life expectancy <24 hours
3. Admitting diagnosis that affects the central nervous system
4. Any reason that the subject may not be able to participate in the follow up assessments (i.e. limb amputation, paresis, neuromuscular disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be enrolling consecutive patients meeting eligibility criteria from each site in this multi-centred study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Regional cerebral oxygenation (rSO2) and delirium | 30 days
  Multivariate linear regression will be used to characterize the association between poor cerebral perfusion (as measured using duration of time (minutes) outside of MAPOPT, mean rSO2, and duration of disturbed cerebral autoregulation) and delirium severity to determine if poor cerebral perfusion is an independent predictor of delirium severity. We will estimate the unadjusted effect of each individual predictor on delirium severity (i.e., cumulative CAM-7 scores per patient). The simultaneous multivariate regression model will adjust for the following covariates (sex, a history of hypertension, a history of alcohol abuse, total sedative dose (in midazolam equivalents), total narcotic dose (fentanyl equivalents), severity of illness (APACHE II scores), pre-existing cognitive impairment (CDR score), length of ICU stay, and blood urea nitrogen. The multivariable model will provide the adjusted regression coefficients after controlling for all predictors included in the model.

SECONDARY OUTCOMES:
Assessment of secondary outcomes-physiological determinants of cerebral oxygenation | 72 hours
  To assess the physiological determinants of rSO2, multiple linear regression will be performed using the patient average of each variable over the 72 hour data collection period. The following predictors will be included in the regression model: heart rate (HR), arterial oxygen saturation (SpO2), MAP, arterial blood gas data (i.e., pH, partial pressure of oxygen, and partial pressure of carbon dioxide), central venous oxygen saturation, and hemoglobin concentration (Hb). In addition, the multivariate model will control for the following covariates associated with cerebral perfusion: sex, age, as well as total sedative, narcotic, and vasopressor dosing. Simultaneous multiple linear regression with adjustment for all aforementioned covariates will be implemented. A within patient repeated measures analysis will also be performed by using the linear mixed effects model with 6 observations per subject reflecting each 12 hour period during the 72 hour data collection period.
Cerebral oxygenation as an independent risk factor for long-term cognitive impairment-RBANS | 3 months and 12 months
  Multiple linear regression analysis will be used to assess if poor cerebral perfusion (i.e. time below MAPOPT, mean rSO2, duration of disturbed cerebral autoregulation) is associated with RBANS global cognition scores at 3- and 12-months post-ICU discharge. We will use the following clinical covariates collected on admission (i.e., pre-existing cognitive impairment, age, severity of illness) and data collected within the first 72 hours of the patients' ICU stay (i.e., narcotic dosing and benzodiazepine dosing). All covariates will be adjusted for in separate regression models for the cognitive outcomes at 3- and 12-months post-ICU discharge. If global cognition is significantly predicted by the impaired cerebral perfusion, we will conduct an exploratory analysis of the RBANS subdomains of cognition (i.e., delay and immediate memory, language, attention, visuospatial/constructional) adjusting for the aforementioned covariates to further explore specific domains of impairment.

OTHER OUTCOMES:
Time outside optimal MAP | 72h, 3- and 12-months
  We define the optimal MAP as the MAP at which there is no statistically significant correlation between MAP and rSO2. The time outside the optimal MAP will be calculated, and will be assessed as an independent predictor of delirium, and 3- and 12-month cognitive outcomes.
Robotic quantification of neurological recovery | 3 and 12 months
  A the Kingston site, participants will undergo additional neurological assessments with the KINARM robot and associated tasks. This data will be analyzed descriptively

CONTACTS AND LOCATIONS:
Overall Officials: J. Gordon Boyd, MD, PhD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khan JM, Wood MD, Lee KFH, Maslove D, Muscedere J, English SW, Ball I, Slessarev M, Boyd JG. Delirium, Cerebral Perfusion, and High-Frequency Vital-Sign Monitoring in the Critically Ill. The CONFOCAL-2 Feasibility Study. Ann Am Thorac Soc. 2021 Jan;18(1):112-121. doi: 10.1513/AnnalsATS.202002-093OC. PMID 32780600
- [Derived] Wood MD, Khan J, Lee KFH, Maslove DM, Muscedere J, Hunt M, Scott SH, Day A, Jacobson JA, Ball I, Slessarev M, O'Regan N, English SW, McCredie V, Chasse M, Griesdale D, Boyd JG. Assessing the relationship between near-infrared spectroscopy-derived regional cerebral oxygenation and neurological dysfunction in critically ill adults: a prospective observational multicentre protocol, on behalf of the Canadian Critical Care Trials Group. BMJ Open. 2019 Jun 25;9(6):e029189. doi: 10.1136/bmjopen-2019-029189. PMID 31243036